CLINICAL TRIAL: NCT07093476
Title: A Multicenter, Randomized, Double-Blind, Placebo-Controlled, Phase 3 Clinical Trial and Open-Label Extension Study to Evaluate the Efficacy and Safety of Add-On Therapy With Empagliflozin for Patients With Inadequately Controlled Type 2 DiabetesMellitus in the Combination Treatment With Metformin and Alogliptin
Brief Title: Efficacy and Safety of Add-On Therapy With Empagliflozin in Patients With Type 2 Diabetes on a Background of Alogliptin and Metformin
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Celltrion (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CT-L02-301
Record Dates: First submitted 2025-06-30; First posted 2025-07-30 (Actual); Last update posted 2025-08-11 (Actual); Status verified 2025-08

CONDITIONS: T2DM; Diabete Type 2; DM
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Metformin; alogliptin; empagliflozin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Study group 1 (Active Comparator): Metformin + Alogliptin + Empagliflozin Xmg
  Interventions: Drug: Metformin; Drug: Alogliptin; Drug: empagliflozin
- Study group 2 (Active Comparator): Metformin + Alogliptin + Empagliflozin Ymg
  Interventions: Drug: Metformin; Drug: Alogliptin; Drug: empagliflozin
- Control Group (Placebo Comparator): Metformin + Alogliptin
  Interventions: Drug: Metformin; Drug: Alogliptin

INTERVENTIONS:
Drug: Metformin — tablets, QD, oral administration
Drug: Alogliptin — tablets, QD, oral administration
Drug: empagliflozin — tablets, QD, oral administration
  Arms: Study group 1; Study group 2

SUMMARY:
Phase 3 study to assess the Efficacy and Safety of CT-L02-301 in Type 2 Diabetes Patients with Insufficient Glycemic Control with Metformin and Alogliptin Combination Therapy.

ELIGIBILITY:
Inclusion Criteria:

* Adults at the time of signing the Informed Consent Form (ICF)
* Signed the written ICF voluntarily after being fully informed of the objectives, methods, and effects of the study
* Diagnosed with T2DM

Exclusion Criteria:

* Diagnosed with other types of diabetes than T2DM
* History of hypersensitivity reaction to the components or drugs of the same class as the IP or the background therapy
* Uncontrolled severe complications of diabetes

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 171 (Estimated)
Dates: Start 2025-07-18 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2027-04 (Estimated)

PRIMARY OUTCOMES:
HbA1c | Week 24 of the Treatment
  Change from Baseline in HbA1c

CONTACTS AND LOCATIONS:
Locations (1):
- Celltrion, Seoul, South Korea